CLINICAL TRIAL: NCT03469557
Title: A Phase 2, Multi-Cohort Study to Investigate the Safety, Pharmacokinetics and Preliminary Antitumor Activity of the Anti-PD-1 Monoclonal Antibody BGB A317 in Combination With Chemotherapy as First-Line Treatment in Adults With Inoperable, Locally Advanced or Metastatic Esophageal, Gastric, or Gastroesophageal Junction Carcinoma
Brief Title: BGB A317 in Combination With Chemotherapy as First-Line Treatment in Adults With Inoperable, Locally Advanced or Metastatic Esophageal, Gastric, or Gastroesophageal Junction Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-205; CTR20170515 (Registry Identifier: ChiCTR)
Record Dates: First submitted 2018-02-08; First posted 2018-03-19 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Esophageal Squamous Cell Carcinoma, Gastric Carcinoma, Gastroesophageal Junction Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Stomach Neoplasms | interventions — tislelizumab; Cisplatin; Fluorouracil; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esophageal Squamous Cell Carcinoma (ESCC) (Experimental)
  Interventions: Drug: Tislelizumab; Drug: Cisplatin; Drug: 5-FU
- Gastric (GC) and Gastroesophageal Junction (GEJ) Carcinoma (Experimental)
  Interventions: Drug: Tislelizumab; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Tislelizumab — Subjects will be treated with BGB A317 200 mg IV on Day 1 during each 21-day cycle. BGB A317 will be administered until disease progression, intolerable toxicity, or treatment discontinuation for any other reason.
  Other Names: BGB-A317
Drug: Cisplatin — Subjects will be treated with cisplatin 80 mg/m² IV on Day 1 during each 21-day cycle. Cisplatinwill be given for up to 6 cycles.
  Arms: Esophageal Squamous Cell Carcinoma (ESCC)
Drug: 5-FU — Subjects will be treated with 5-FU 800 mg/m²/day IV using continuous pumping system on Days 1 through 5 during each 21-day cycle. 5-FU will be given for up to 6 cycles.
  Arms: Esophageal Squamous Cell Carcinoma (ESCC)
Drug: Oxaliplatin — Subjects will be treated with oxaliplatin 130 mg/m² IV on Day 1 during each 21-day cycle. Oxaliplatin will be administered for up to 6 cycles.
  Arms: Gastric (GC) and Gastroesophageal Junction (GEJ) Carcinoma
Drug: Capecitabine — Subjects will be treated with capecitabine 1000 mg/m² orally twice daily (bid) Days 1 through 14 (14 days total) during each 21-day cycle. Capecitabine will be administered until disease progression, intolerable toxicity, or treatment discontinuation for any other reason.
  Arms: Gastric (GC) and Gastroesophageal Junction (GEJ) Carcinoma

SUMMARY:
This is a Phase 2, multi-cohort study to investigate safety, PK, and preliminary anti-tumor activity of the monoclonal antibody BGB A317 in combination with standard chemotherapy as first-line treatment. Cohorts include an ESCC cohort and a gastric carcinoma (GC) or GEJ carcinoma cohort that will be enrolled concurrently. The study includes a screening (up to 28 days), treatment (until disease progression, intolerable toxicity, or treatment withdrawal for another reason), safety follow-up (up to 30 days following last study drug treatment), and survival follow-up phase.

DETAILED DESCRIPTION:
The study includes an initial phase during which 6 subjects will be enrolled in each cohort (ESCC and GC/GEJ carcinoma). Safety data will be reviewed by a Safety Monitoring Committee (SMC) after the first 6 subjects in a cohort have completed at least 1 cycle (21 days) of treatment. During the initial phase, subjects who discontinue for a reason unrelated to safety before completing Cycle 1 will be replaced. If there are no new, significant or severe, safety signals detected, the enrollment will be expanded up to approximately 15 subjects per cohort (treatment expansion). During the treatment expansion, subjects will not be replaced for any reason.

In the ESCC cohort, subjects will be treated with BGB A317 200 mg IV on Day 1, cisplatin 80 mg/m² IV on Day 1, and 5-FU 800 mg/m²/day IV using continuous pumping system on Days 1 through 5 during each 21-day cycle. Cisplatin and 5-FU will be given for up to 6 cycles and BGB A317 will be administered until disease progression, intolerable toxicity, or treatment discontinuation for any other reason.

In the GC and GEJ carcinoma cohort, subjects will be treated with BGB A317 200 mg IV on Day 1, oxaliplatin 130 mg/m² IV on Day 1, and capecitabine 1000 mg/m² orally twice daily (bid) Days 1 through 14 (14 days total) during each 21-day cycle. Oxaliplatin will be administered for up to 6 cycles and capecitabine and BGB A317 will be administered until disease progression, intolerable toxicity, or treatment discontinuation for any other reason.

ELIGIBILITY:
Key Inclusion Criteria:

1. Pathologically (histologically or cytologically) confirmed diagnosis of either inoperable, locally advanced or metastatic gastric/GEJ adenocarcinoma that is HER2/neu negative or inoperable, locally advanced or metastatic ESCC.

   Note: Archival tumor tissue (paraffin blocks or at least 10 unstained tumor specimen slides) must be available for biomarker analysis. In the absence of archival tumor tissues, a fresh biopsy of a tumor lesion at baseline is mandatory. Subjects may be permitted to enroll on a case-by-case basis after discussion with the Sponsor's medical monitors if paraffin block is not available and fewer than 10 unstained slides can be provided.
2. Have received no prior systemic therapy for advanced or metastatic disease. Subject may have received prior neoadjuvant or adjuvant therapy provided it was completed at least 6 months prior to enrollment.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (Protocol Appendix 3).
4. Life expectancy of at least 12 weeks.
5. Adequate organ function as indicated by the following screening laboratory values:

Absolute neutrophil count (ANC) ≥1.5×109/L Platelet count ≥100×109/L Hemoglobin ≥9 g/dL or ≥5.6 mmol/L (Note: Criteria must be met without a transfusion within 4 weeks before sample is drawn).

Serum creatinine ≤1.5× upper limit of normal (ULN). Serum total bilirubin ≤1.5×ULN. For subjects with Gilbert's syndrome, total bilirubin must be <3×ULN) Prothrombin time/international normalized ratio (PT/INR) ≤1.5×ULN and activated partial thromboplastin time (aPTT) ≤1.5×ULN unless subject is receiving anticoagulant therapy and PT values is within the intended therapeutic range of the anticoagulant.

Aspartate transaminase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN. For subjects with liver metastases, AST and ALT must be ≤5×ULN for subjects with liver metastases

Key Exclusion Criteria:

1. History of severe hypersensitivity reactions to other mAbs; has known hypersensitivity to fluorouracil (5-FU), cisplatin, or other platinum agents
2. Unable to receive a port or peripherally inserted central catheter (PICC) for ESCC subjects
3. Prior malignancy active within the 2 years prior to Cycle 1 Day 1, exceptions include the tumor under investigation in this study, and locally recurring cancers that have undergone curative intent treatment, such as resected basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix or breast.
4. Received prior therapies targeting PD-1, PD-L1 or PD-L2 for any reason.
5. Have known active brain or leptomeningeal metastases. Subjects with brain metastases are permitted if they are asymptomatic or had previously treated brain metastases that are asymptomatic, radiographically stable and did not require steroid medications for at least 4 weeks prior to Cycle 1 Day 1
6. Active autoimmune diseases or history of autoimmune diseases that may relapse should be excluded (Protocol Appendix 5). Subjects with following diseases are allowed to undergo screening: type I diabetes, hypothyroidism managed with hormone replacement therapy only, skin diseases not requiring systemic treatment (such as vitiligo, psoriasis or alopecia), controlled celiac disease, or diseases not expected to recur in the absence of external triggering factors.
7. Requires systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration to treat a current condition.

   Note:Adrenal replacement doses ≤10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease; subjects are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
8. History of interstitial lung disease, non-infectious pneumonitis except for those induced by radiation therapies; uncontrolled systemic diseases, including diabetes, hypertension, pulmonary fibrosis, acute lung diseases, etc.
9. Severe chronic or active infection requiring systemic antibacterial, antifungal or antiviral therapy, including tuberculosis infection, etc.
10. Uncontrollable pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
11. Any of the following cardiovascular criteria:

    * Current evidence of cardiac ischemia
    * Current symptomatic pulmonary embolism
    * Acute myocardial infarction ≤6 months prior to Day 1
    * Heart failure of New York Heart Association Classification III or IV(Protocol Appendix 6) ≤6 months prior to Day 1
    * Grade 2 or higher ventricular arrhythmia ≤6 months prior to Day 1
    * Cerebral vascular accident (CVA) or transient ischemic attack (TIA) ≤6 months prior to Day 1
12. Has a history of alcohol or drug abuse or dependence
13. Known history of Human Immunodeficiency Virus (HIV).
14. Untreated chronic hepatitis B viral (HBV) infection or chronic HBV carrier with HBV DNA ≥200 IU/mL (or 1000 copies/mL), or active hepatitis C virus (HCV) should be excluded. Note: subjects with inactive HBV surface antigen (HBsAg) carrier, active HBV infection with sustained anti-HBV suppression (HBV DNA <200 IU/mL or 1000 cps/mL), and subjects whose HCV has been cured can be enrolled.
15. Underlying medical conditions that, in the investigator's opinion, will be unfavorable for the administration of study drug or affect communication regarding drug toxicity or adverse events. Note: subjects whose compliance during this study is considered by the investigator to be questionable should be excluded.
16. Has been administered a live vaccine within 4 weeks prior to Cycle1 Day 1.
17. Administered a monoclonal antibody within 4 weeks for any reason prior to study Day 1 or who has not recovered (i.e., Grade 1 or lower at baseline) from adverse events due to agents administered more than 4 weeks earlierMedical history of dihydropyrimidine dehydrogenase deficiency (DPD). Note: subjects do not need to be tested for DPD at screening.
18. Medical history of dihydropyrimidine dehydrogenase deficiency (DPD). Note: subjects do not need to be tested for DPD at screening.
19. Has received radiotherapy or treatment with an investigational agent within 14 days prior to Cycle 1 Day 1
20. Major surgical procedure other than for diagnostic biopsy of tumor tissue for this study or placement of a venous access device within 28 days prior to study drug administration.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2020-08-19 (Actual)

PRIMARY OUTCOMES:
The objective response rate (ORR) as assessed by RECIST, Version 1.1 | Through study completion, an average of 9 months
The Duration of Response (DoR) as assessed by RECIST, Version 1.1 | Through study completion, an average of 9 months
The Disease Control Rate (DCR) as assessed by RECIST, Version 1.1 | Through study completion, an average of 9 months
The Progression-Free Survival (PFS) as assessed by RECIST, Version 1.1 | Through study completion, an average of 9 months
Pharmacokinetic evaluations: include but not limited to minimum observed serum concentration (Ctrough) for BGB-A317. | Through study completion, an average of 10 months
Host immunogenicity: BGB-A317 anti-drug antibody (ADA) | Through study completion, an average of 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Xu, MD, Principal Investigator — The fifth Medical Center, Chinese PLA General Hospital
Locations (6):
- China (6):
  - Fifth Medical Center of Pla General Hospital, Beijing, Beijing Municipality
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Northern Jiangsu Peoples Hospital, Yangzhou, Jiangsu
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Upon request, and subject to certain criteria, conditions, and exceptions, BeiGene will provide access to individual de-identified participant data from BeiGene-sponsored global interventional clinical studies conducted for medicines for indications that have been approved or in programmes that have been terminated. BeiGene will also consider requests for the protocol, data dictionary, and statistical analysis plan. Data requests can be submitted to medicalinformation@beigene.com.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Xu J, Bai Y, Xu N, Li E, Wang B, Wang J, Li X, Wang X, Yuan X. Tislelizumab Plus Chemotherapy as First-line Treatment for Advanced Esophageal Squamous Cell Carcinoma and Gastric/Gastroesophageal Junction Adenocarcinoma. Clin Cancer Res. 2020 Sep 1;26(17):4542-4550. doi: 10.1158/1078-0432.CCR-19-3561. Epub 2020 Jun 19. PMID 32561664